CLINICAL TRIAL: NCT01853527
Title: Myocardial Ischemia in Non-obstructive Coronary Artery Disease
Acronym: MicroCAD
Status: Completed | Type: Observational
Sponsor: University of Bergen (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Mai Tone Lønnebakken, MD, phd, University of Bergen
Other Study IDs: 2012/2167b
Record Dates: First submitted 2013-05-07; First posted 2013-05-15 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Coronary Atherosclerosis; Myocardial Ischemia
Keywords: CT coronary angiography; Contrast stress echocardiography; Arterial stiffness; Quality of life; Biochemical and genetic markers
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urin test for biobank
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Angina pectoris, non-obstructive CAD: Contrast stress echocardiography will be performed in patients with angina pectoris and non-obstructive CAD on CT-angiography to detect presence of myocardial ischemia

SUMMARY:
The aim of the study is to assess presence of myocardial ischemia by contrast stress echocardiography in patients with symptomatic non-obstructive coronary artery disease (CAD) by CT-coronary angiography, and the clinical, vascular, biochemical and genetic markers of myocardial ischemia in such patients.

DETAILED DESCRIPTION:
Non-obstructive coronary artery disease (CAD) is particularly common in women and associated with reduced quality of life and increased cardiovascular morbidity and mortality. The project will recruit patients with angina pectoris and non-obstructive CAD by CT- coronary angiography for further imaging with contrast stress echocardiography for diagnosis of myocardial ischemia. Better characterization of patients with symptomatic non-obstructive CAD due to myocardial ischemia will be done by vascular assessment by tonometry, biochemical and genetic markers as well as quality of life questionnaire. This interdisciplinary project is expected to add new knowledge to the impact of multimodality cardiac imaging in improving diagnosis in patients with symptomatic non-obstructive CAD.

ELIGIBILITY:
Inclusion Criteria:

* Age >30 years
* Chest pain and or functional dyspnoea with a duration > 6 months
* Non-obstructive coronary artery disease detected by CT coronary angiography

Exclusion Criteria:

* Significant coronary artery stenosis or normal coronary arteries by CT coronary angiography
* Unstable coronary artery disease
* Significant valvular heart disease
* Mechanical valve prosthesis
* Significant arrhythmia
* Severly reduced pulmonary function (GOLD 3-4)
* Known allergy to ultrasound contrast agents
* Pregnancy
* Inability to sign informed consent to participate
* Other severe disease

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population include 132 patients with symptomatic angina pectoris and non-obstructive coronary artery disease detected by CT-coronary angiography
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2013-04; Primary Completion 2015-05 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Presence of myocardial ischemia by contrast stress echocardiography | 15 minutes, during contrast stress echocardopgraphy
  Presence of delayed myocardial contrast enhancement during stress echocardiography

SECONDARY OUTCOMES:
Extent of myocardial ischemia by contrast stress echocardiography | 15 minutes, during contrast stress echocardiography
  Numbers of left ventricular segments with delayed contrast enhancement during stress echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Mai Tone Lønnebakken, MD, phd, Principal Investigator — University of Bergen
Locations (1):
- Department of Heart Disease, Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Derived] Eskerud I, Gerdts E, Larsen TH, Simon J, Maurovich-Horvat P, Lonnebakken MT. Total coronary atherosclerotic plaque burden is associated with myocardial ischemia in non-obstructive coronary artery disease. Int J Cardiol Heart Vasc. 2021 Jun 30;35:100831. doi: 10.1016/j.ijcha.2021.100831. eCollection 2021 Aug. PMID 34258383
- [Derived] Lonnebakken MT, Eskerud I, Larsen TH, Midtbo HB, Kokorina MV, Gerdts E. Impact of aortic stiffness on myocardial ischaemia in non-obstructive coronary artery disease. Open Heart. 2019 May 4;6(1):e000981. doi: 10.1136/openhrt-2018-000981. eCollection 2019. PMID 31217997